CLINICAL TRIAL: NCT02390284
Title: Stop Retinal Ganglion Cell Dysfunction Study
Acronym: STOP-RGCD
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: No patients had abnormal PERG and could not be included in the first two arms from the baseline timepoint.
Sponsor: University of Miami (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Vittorio Porciatti, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20140587; R01EY014957 (NIH)
Record Dates: First submitted 2015-03-10; First posted 2015-03-17 (Estimated); Results first posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Glaucoma
Keywords: RGCD; Glaucoma Suspect
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — Latanoprost; Bimatoprost; Travoprost; Timolol; dorzolamide; brinzolamide; Acetazolamide; Methazolamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Abnormal PERG Untreated (No Intervention): Participants recognized as Glaucoma suspects with an abnormal PERG test who have been assigned to not receive therapy or intervention.
- Abnormal PERG Treated (Experimental): Participants recognized as Glaucoma suspects with an abnormal PERG test who have been assigned to receive one or more drops in each eye in order to reduce the intraocular pressure by 20%.
  Drugs could be:
  Latanoprost 1 drop Once a day (QD) Bimatoprost 1 drop QD Travoprost 1 drop QD Timolol 1 drop Twice a day (BID) Dorzolamide 1 drop Three times a day (TID) Brinzolamide 1 drop BID Acetazolamide and Methazolamide depends on clinicians evaluation.
  If Clinicians consider necessary, he/she might combine 2 drugs in order to get the desired intraocular pressure.
  Interventions: Drug: Latanoprost; Drug: Bimatoprost; Drug: Travoprost; Drug: Timolol; Drug: Dorzolamide; Drug: Brinzolamide; Drug: Acetazolamide; Drug: Methazolamide
- Normal (No Intervention): Patients with a normal PERG test that will go through the study under observation.

INTERVENTIONS:
Drug: Latanoprost — Lower intraocular pressure (IOP) by increasing outflow of fluid from the eye.
  Other Names: Xalatan
  Arms: Abnormal PERG Treated
Drug: Bimatoprost — Lower intraocular pressure by increasing outflow of fluid from the eye.
  Other Names: Lumigan
  Arms: Abnormal PERG Treated
Drug: Travoprost — Lower intraocular pressure by increasing outflow of fluid from the eye.
  Other Names: Travatan
  Arms: Abnormal PERG Treated
Drug: Timolol — Lower intraocular pressure by decreasing production of fluid
  Other Names: Timoptic
  Arms: Abnormal PERG Treated
Drug: Dorzolamide — Lowers intraocular pressure by decreasing intraocular fluid production
  Other Names: Trusopt
  Arms: Abnormal PERG Treated
Drug: Brinzolamide — Lowers intraocular pressure by decreasing intraocular fluid production
  Other Names: Azopt
  Arms: Abnormal PERG Treated
Drug: Acetazolamide — Lowers intraocular pressure by decreasing intraocular fluid production
  Other Names: Diamox
  Arms: Abnormal PERG Treated
Drug: Methazolamide — Lowers intraocular pressure by decreasing intraocular fluid production
  Other Names: Neptazane
  Arms: Abnormal PERG Treated

SUMMARY:
Glaucoma is a progressive disease resulting in blindness. Determining the onset of the disease, predicting its severity and the benefit of pressure lowering eye drops is key to clinical management aimed at maintaining useful vision with advancing age. This study will longitudinally monitor a population of glaucoma suspects (with positive factors for the disease but with normal vision) with noninvasive pattern electroretinogram (PERG) and other standard eye tests for glaucoma. The PERG measures the function of retinal ganglion cells (RGCs) that are the parent neurons of the optic nerve. RGCs may become dysfunctional before dying and their function restored with pressure-lowering eye drops. Glaucoma suspects with abnormal PERG will be randomized to treatment with eye drops, while those with normal PERG will be left untreated. All patients will be monitored with PERG, Optic Coherence Tomography (OCT) and other ancillary tests every 6 months over 4 years.

DETAILED DESCRIPTION:
The PERG is recorded from small metallic buttons taped on the skin similarly to an electrocardiogram, with the difference that the electrodes are around the eyes.

The only physical contact you will experience is a gentle cleaning of the skin with an alcohol prep pad. During the test you must look with both eyes at a Television (TV) display for about 3 minutes. During the follow up period you may be asked to take one more PERG test lying down in a bed.

This will cause a momentary increase of your eye pressure similar to the one that occurs during your normal sleep. This may help to understand whether or not your optic nerve functions normally when the pressure in your eye increases. For OCT evaluation, the pupil has to be dilated with drops as you did before for your eye exam. You have to briefly look at a mark inside the instrument one eye at a time.

PERG and OCT will be performed during the same day of your visit with the eye doctor. If you have already done these tests in the past, as part of another study or as part of your standard treatment, the results of these tests will be obtained from your record, and be included in this study.

If you are a participant in the Observation Group, you will be monitored with PERG, OCT, and standard clinical examinations every six months until close of study. If you are a participant in the Medication Group you will be also treated with eye drop medicines.

RISKS:

There are certain risks and discomforts that may be associated with this research. You should be aware that you are at risk of developing glaucoma whether you participate in the study or not. It is not known whether the risk of developing glaucoma is reduced by eye drops to lower eye pressure; the study will attempt to answer this question.

For the PERG, the only significant risk to you is a small chance of a rash to the cleansing agent for skin electrodes, which should go away without treatment. For OCT, there is a rare risk to you of an allergic reaction to the drops used to dilate your pupils. The risk is even lower if you did not have any reaction during your previous eye exams. In case of an allergic reaction, your eye doctor will immediately treat it. If you had previous problems with pupil dilation, you may wish to speak to your eye doctor about the option of doing this additional test.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 85 years, inclusive
2. Refractive errors within -5 to +3 diopters
3. Best corrected visual acuity (BCVA) better than or equal to 20/30 (Snellen)
4. Normal standard automated perimetry (SAP) according to the Ocular Hypertension Treatment Study (OHTS) criteria15 (reliability < 15% on all indices, normality > 5% on all global indices in two consecutive sessions 6 months apart)
5. Minimum untreated Intraocular pressure IOP of 15 mm Hg
6. Glaucoma Suspect Status defined as one or more of the following:

   * Glaucomatous optic disc appearance (vertical cup-to-disc ratio [C/D] ≥0.5
   * Cup disc ratio asymmetry ≥0.2
   * Localized thinning of the disc
   * Presence or history of splinter disc hemorrhage
   * Moderately increased IOP (>21 to <28 mm Hg).
   * Family history of vision loss for glaucoma

Exclusion Criteria:

1. Age-related macular degeneration
2. Diabetes
3. Parkinson's disease
4. Multiple sclerosis
5. Unwilling or unable to give consent, unwilling to accept randomization, or unable to return for scheduled protocol visits.
6. Pregnant or nursing women.
7. Currently using prescribed pressure lowering medicines and unwilling to be withdrawn from them.
8. An OHTS risk score high enough in the judgment of the ophthalmologist or optometrist managing the patient to recommend pressure lowering medicine to the patient and not randomization.
9. An OCT abnormal enough in a pattern consistent with glaucoma.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2024-10-04 (Actual); Study Completion 2024-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vittorio Porciattti, DSc, Principal Investigator — University of Miami
Locations (1):
- Bascom Palmer Eye Institute - University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No patients had abnormal PERG and could not be included in the first two arms from the baseline timepoint. This significantly altered the study since the patients could not be randomized, and the treatment of each patient was determined by the physician's discretion.
Groups:
- Abnormal PERG Treated: Participants recognized as Glaucoma suspects with an abnormal PERG test who have been assigned to receive one or more drops in each eye in order to reduce the intraocular pressure by 20%.
  Drugs could be:
  Latanoprost 1 drop Once a day (QD) Bimatoprost 1 drop QD Travoprost 1 drop QD Timolol 1 drop Twice a day (BID) Dorzolamide 1 drop Three times a day (TID) Brinzolamide 1 drop BID Acetazolamide and Methazolamide depends on clinicians evaluation.
  If Clinicians consider necessary, he/she might combine 2 drugs in order to get the desired intraocular pressure.
  Latanoprost: Lower intraocular pressure (IOP) by increasing outflow of fluid from the eye.
  Bimatoprost: Lower intraocular pressure by increasing outflow of fluid from the eye.
  Travoprost: Lower intraocular pressure by increasing outflow of fluid from the eye.
  Timolol: Lower intraocular pressure by decreasing production of fluid
  Dorzolamide: Lowers intraocular pressure by decreasing intraocular fluid production
  Brinzolamide: Lowers intraocular pressure by decreasing intraocular fluid production
  Acetazolamide: Lowers intraocular pressure by decreasing intraocular fluid production
  Methazolamide: Lowers intraocular pressure by decreasing intraocular fluid production
Period: Overall Study
Arm/Group | Abnormal PERG Untreated | Abnormal PERG Treated | Normal
Started | 0 (No patients had abnormal PERG and could not be included in this arm.) | 0 (No patients had abnormal PERG and could not be included in this arm.) | 28
Completed | 0 (No patients had abnormal PERG and could not be included in this arm.) | 0 (No patients had abnormal PERG and could not be included in this arm.) | 19
Not Completed | 0 | 0 | 9
Not completed — Physician Decision | 0 | 0 | 9

BASELINE CHARACTERISTICS:
Population: No patients had abnormal PERG and could not be included in the first two arms.
Groups:
- Total: Total of all reporting groups
Arm/Group | Abnormal PERG Untreated | Abnormal PERG Treated | Normal | Total
Number analyzed (Participants) | 0 | 0 | 28 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  |  | 0 | 0
  Between 18 and 65 years |  |  | 16 | 16
  >=65 years |  |  | 12 | 12
Age, Continuous [Mean (Full Range); unit: years] |  |  | 62.03 [20 to 81] | 62.03 [20 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  |  | 19 | 19
  Male |  |  | 9 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  |  | 0 | 0
  Asian |  |  | 0 | 0
  Native Hawaiian or Other Pacific Islander |  |  | 0 | 0
  Black or African American |  |  | 4 | 4
  White |  |  | 24 | 24
  More than one race |  |  | 0 | 0
  Unknown or Not Reported |  |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  |  | 28 | 28
PERG Amplitude [Mean (Full Range); unit: nanovolts] |  |  | 787.785714 [274 to 1560] | 787.785714 [274 to 1560]
PERG Phase [Mean (Full Range); unit: degrees] |  |  | 66.92857 [15 to 106] | 66.92857 [15 to 106]
IOP [Mean (Full Range); unit: mmHg] |  |  | 18 [13 to 24] | 18 [13 to 24]
OCT-RNFL thickness [Mean (Full Range); unit: micrometers] |  |  | 85 [76 to 96] | 85 [76 to 96]
Visual Field [Number; unit: participants] — A test in which a patient sees a visual stimulus and pushes a button whenever it appears, this maps the ability to detect areas of visual loss.
  A normal visual field, as measured in decibels (dB) using an Automated Perimetry machine, typically falls within the range of 0 to -2 dB, specifically referring to the Mean Deviation (MD) value. Values more negative than -2 dB indicate visual field loss.
  The standard automated analysis is able to classify tests as "Within Normal Limits" or "Abnormal", here we measured the number of subjects that classified as "Within Normal Limits".
  participants |  |  | 28 | 28

OUTCOME MEASURES:

1. Primary Outcome: Retinal Nerve Fiber Layer Thickness
Description: As measured by Optical Coherence Tomography in different timepoints as an absolute value in micrometers.
Time Frame: Baseline
Population: No patients had abnormal PERG and could not be included in the first two arms from the baseline timepoint, only baseline measurements could be included.
Measure: Mean (Full Range); unit: micrometers
Arm/Group | Abnormal PERG Untreated | Abnormal PERG Treated | Normal
Number analyzed (Participants) | 0 | 0 | 28
micrometers |  |  | 79 [76 to 89]

2. Secondary Outcome: Pattern Electroretinogram Amplitude
Description: Assessed via Pattern Electroretinogram in nanovolts
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Full Range); unit: nanovolts
Arm/Group | Abnormal PERG Untreated | Abnormal PERG Treated | Normal
Number analyzed (Participants) | 0 | 0 | 28
nanovolts |  |  | 706 [455 to 1344]

3. Secondary Outcome: Pattern Electroretinogram Phase
Description: Assessed via Pattern Electroretinogram in degrees
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Full Range); unit: degrees
Arm/Group | Abnormal PERG Untreated | Abnormal PERG Treated | Normal
Number analyzed (Participants) | 0 | 0 | 28
degrees |  |  | 67.34 [22 to 96]

ADVERSE EVENTS:
Time Frame: 4 years
Arm/Group | Abnormal PERG Untreated | Abnormal PERG Treated | Normal
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/28
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/28

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed and qualifying for the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-10-30): https://cdn.clinicaltrials.gov/large-docs/84/NCT02390284/Prot_SAP_000.pdf
  • Informed Consent Form (2019-05-13): https://cdn.clinicaltrials.gov/large-docs/84/NCT02390284/ICF_001.pdf